CLINICAL TRIAL: NCT05475964
Title: Assistant Lecturer of Tropical Medicine and Gastroenterology
Brief Title: The Role of Endoscopic Ultrasound in Evaluation of Patients With Indefinite Cause of Bile Duct Dilatation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: HMHamed (Other)
Responsible Party: Sponsor-Investigator, HMHamed, Assistant lecturer of tropical medicine and gastroenterology, Assiut University
Organization: Assiut University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EUS in biliary dilatation
Record Dates: First submitted 2022-07-20; First posted 2022-07-27 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Bile Duct Diseases
MeSH Terms: conditions — Bile Duct Diseases | interventions — Endosonography

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients with undiagnosed bile duct dilatation (Other): patients with bile duct dilation detected by imaging studies without revealing definite cause of obstruction
  Interventions: Device: Endoscopic ultrasound

INTERVENTIONS:
Device: Endoscopic ultrasound — Endoscopic ultrasound and biopsy intake of suspected lesions

SUMMARY:
In the era of diagnostic imaging advances, Bile Duct Dilatation becomes a common incidental finding in patients present with either gastrointestinal symptoms or undergone the imaging study for any other complaints. Endoscopic ultrasound enables high resolution views of the biliary system, so it can help detection of different pathologies which cause bile duct dilatation and difficult to be detected by other imaging studies.

DETAILED DESCRIPTION:
The normal diameter of the common bile duct (CBD) varies by age, imaging modality, prior cholecystectomy, and previous biliary obstruction, but 7 mm or more is considered widely accepted cutoff for biliary dilatation, and 10 mm or more among post-cholecystectomy patients.

BDD with unclear etiology detected on trans abdominal ultrasound (TUS), computed tomography (CT), or magnetic resonance cholangiopancreatography (MRCP). Although, these imaging techniques have a good sensitivity and specificity in detecting biliary tract diseases, limitations are still present in the detection of intraductal small stones, ampullary lesions and small masses.

As regard TUS, overlying bowel gas and operator-dependence, often harshen an adequate visualization of the biliary duct to identify the etiology, and CT could miss tumors less than 2 cm in size, while the sensitivity of MRCP decreases in stones 3 mm or less in size.

Endoscopic ultrasound (EUS) enables high resolution views of the biliary tree as it joins the pancreatic duct and duodenum, so it helps detection of biliary pathologies difficult to be diagnosed by external radiograph. In addition, EUS is less invasive than the competitive endoscopic retrograde cholangiopancreatography (ERCP) as a diagnostic modality and it avoids the patients the post-ERCP pancreatitis which is a very common complication, as well as providing a unique opportunity of tissue sampling and staging of any detected malignant lesions.

Previously, EUS has proven it's high ability to the detect the stones in the extrahepatic ducts with a sensitivity as high as of 94% and specificity of 95%.

Besides, it's well performance in the evaluation of biliary strictures with a sensitivity 80%, and a specificity of 97% in detecting malignant biliary strictures.

When it comes to ampullary and pancreatic lesions, direct endoscopic visualization with a side-viewing endoscope can effectively evaluate the periampullary area and detect ampullary mass and diverticulum, as well examine the pancreas for chronic pancreatitis, masses, and cysts.

ELIGIBILITY:
Inclusion Criteria:

1. Prior inconclusive imaging studies of bile duct dilation.
2. Common bile duct diameter of >10 mm with prior cholecystectomy or >7 mm without

Exclusion Criteria:

Definite cause of obstruction stone, stricture, or mass on imaging studies (TUS, CT, MRCP or ERCP).

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-09-09 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
The percentage of patients with bile duct dilatation | 2 years
  Can EUS detect the cause of bile duct dilatation in patients not diagnosed by other imaging modalities

CONTACTS AND LOCATIONS:
Overall Officials: Hager Hamed, Master, Principal Investigator — Assiut University
Locations (1):
- AssiutU, Asyut, Egypt